CLINICAL TRIAL: NCT02243865
Title: A Randomized, Placebo-controlled, Double-blind, Multi-center Clinical Investigation to Evaluate the Prophylactic Effect and Tolerability of Intranasal Kinetic Oscillation Stimulation (KOS) Using the Chordate System S200 in Migraine Patients
Brief Title: Chordate System Prophylactic Migraine Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chordate Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PM005
Record Dates: First submitted 2014-09-10; First posted 2014-09-18 (Estimated); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A placebo module, with one input and 6 outputs, was added to the Chordate S200 system. Some outputs delivered active treatment and others placebo. The operator received a coded envelope and according to that, either active treatment or placebo was selected. The operator did not know which outputs delivered treatment and which did not.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chordate S200 + control module (CT100), active (Experimental): Chordate System S200 giving Kinetic Oscillation Stimulation Treatment for 15 minutes in each nostril
  Interventions: Device: Chordate System S200 + CT100 (active treatment)
- Chordate S200 + control module (CT100), placebo (Placebo Comparator): Chordate System S200 giving Kinetic Oscillation Stimulation in placebo mode. Non-inflated and non-vibrating treatment
  Interventions: Device: Chordate System S200 + CT100 (placebo treatment)

INTERVENTIONS:
Device: Chordate System S200 + CT100 (active treatment) — Chordate S200 + CT100 (active treatment) gives Kinetic Oscillation Stimulation for 15 minutes to each nostril and by that giving an effect on the autonomic nervous system (ANS).
  Arms: Chordate S200 + control module (CT100), active
Device: Chordate System S200 + CT100 (placebo treatment) — Chordate S200 + CT100 (placebo) is used in the same way as Active treatment, but no Kinetic Oscillation Stimulation is given. Catheter is not inflated and no vibration is given.
  Arms: Chordate S200 + control module (CT100), placebo

SUMMARY:
The purpose of this pilot study is to evaluate the performance of the Chordate System, in terms of the prophylactic effect and tolerability of treatment in patients diagnosed with migraine.

DETAILED DESCRIPTION:
This was a prospective, interventional, randomized, placebo-controlled, double-blind, multi-center clinical investigation of a medical device system.

A pilot study in which patients with frequent migraine attacks received intranasal KOS or placebo using the Chordate System S200 on two occasions.

ELIGIBILITY:
Inclusion Criteria:

* The subject is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the Informed Consent Form (ICF).
* Male or female aged between 18 and 65 years
* Diagnosed as suffering from migraine with or without aura according to International Headache Society´s (IHS) classification (International Classification of Headache Disorders (ICHD), 3rd edition, beta version)
* Reported history of 3 to 8 migraine episodes per month during previous 2 months, confirmed during baseline
* Reported history of at least 48 hours of freedom from headache between migraine attacks, confirmed during baseline
* Onset of migraine headache occurred before age 50
* Reported history of migraine for more than one year
* Reported stable dose of prophylactic migraine medication(s), if any, during the two months prior to screening (visit 1), and willing and able to maintain stable dose(s) until the three months follow-up (visit 4)

Exclusion Criteria:

* Meeting the ICHD criteria for medication overuse
* Reported history of 15 or more headache days per month (i.e. headaches of any kind), confirmed during baseline
* Reported frequency of non-migraine headaches exceeding 6 days per month, confirmed during baseline
* Unable to distinguish between migraine headaches and other headache types
* Treatment with Botox received within 6 months of the screening visit, or between the screening and treatment visits
* Ongoing treatment with implanted stimulator or other implanted device in the head and/or neck region
* Known pronounced anterior septal deviation, or other known relevant abnormality in the nasal cavity, including bacterial infection and wounds
* History of sinus surgery, transphenoidal surgery for pituitary or other lesions or cerebrospinal fluid (CSF) rhinorrhea
* Fitted with a pacemaker/defibrillator
* Previously treated with therapeutic radiation to the face (that could have influenced the nasal mucosa)
* Ongoing upper respiratory tract infection or a body temperature >38.5°C (at treatment), or malignancy in the nasal cavity
* History of regular nose bleeding (epistaxis), or concomitant condition that could cause excessive bleeding, including treatment with the anticoagulant Varan
* Head injury or open wound that contraindicates use of Chordate Headband
* Known allergy to polyvinylchloride, a material used in the Catheter, or medicinal liquid paraffin
* Concurrent condition or risk of non-compliance that, in the investigator's opinion, may affect the interpretation of performance or safety data or which otherwise contraindicates participation in a clinical investigation
* Any change in migraine prophylaxis the previous two months
* Pregnant women
* Participation in a clinical research study within three months of enrolment or planned participation at any time during this clinical investigation
* Employees of the study site or the sponsor directly involved with the conduct of the study, or immediate family members or any such individuals
* Headache or migraine episode within the 48 hours prior to the first treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Åke Åkesson, MD, Study Chair — Linkoeping University
Locations (4):
- Sweden (4):
  - Stortorgets neurologmottagning, Helsingborg
  - Läkarcentrum Stångåblick, Linköping
  - Neurolgy Clinic, Stockholm
  - Neurologmottagningen Vällingby sjukhus, Vällingby

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Chordate System S200 + CT100 (Active) Treatment: Chordate System S200 + control module (CT100), active treatment: 44 subjects
- Chordate System S200 + CT100 (Placebo Treatment): Chordate System S200 + control module (CT100), placebo treatment: 38 subjects
Period: Overall Study
Arm/Group | Chordate System S200 + CT100 (Active) Treatment | Chordate System S200 + CT100 (Placebo Treatment)
Started | 44 | 43
Completed | 40 | 38
Not Completed | 4 | 5
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Chordate System S200 + CT100 (Active Treatment): Chordate System S200 + CT100 (active treatment) is Kinetic Oscillation Stimulation (KOS) treatment with the Chordate System S200 + CT100
- Chordate System S200 + CT100 (Placebo Treatment): Chordate System S200 + CT100 (placebo treatment), is Placebo treatment with the Chordate System S200 + CT100 without an inflated catheter and without vibrations
- Total: Total of all reporting groups
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment) | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 43 | 87
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (11.7) | 49.0 (10.5) | 47.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  Sweden | 44 | 43 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Migraine Days Per Four Weeks During the Three Months Post Treatment Investigation Duration
Description: A diary was used where patients added information each day on experienced migraine (yes/no). Baseline was defined as any migraine days from Day -29 until Day -1, i.e. the day before first treatment (Day 1). If full time period for baseline or the post treatment period was not documented, number of migraine days was recalculated with the formula:
  Number of migraine days = (Number of migraine days x 28) / Number of days observed
  If data was missing for any patient for more than 14 days during any period of interest, that patient was excluded from analysis.
  The change from baseline in number of migraine days was calculated as follows:
  Change = number of migraine days per four weeks for the 3 months post treatment period - number of migraine days per four weeks of the baseline period
  As the difference between the post treatment period and baseline is presented, negative numbers indicate a post treatment decrease in number of migraine days.
Time Frame: From baseline (28 days pre-treatment) to visit 4 (day 98, ± 7 days)
Population: 44 patients were allocated to active treatment and 43 to placebo. Out of these 40 patients completed the active treatment and 38 patients completed placebo treatment. Only patients who completed treatment were included in analysis (see participant flow).
Measure: Mean (Standard Deviation); unit: Migraine days/four weeks
Groups:
- Chordate System S200 + CT100 (Active Treatment): Chordate System S200 + CT100 (active treatment): 44 subjects
- Chordate System S200 + CT100 (Placebo Treatment): Chordate System S200 + CT100 (placebo treatment): 43 subjects
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment)
Number analyzed (Participants) | 40 | 38
Migraine days/four weeks | -1.5 (3.6) | -1.3 (3.0)
Statistical Analysis 1: Comparison: Chordate System S200 + CT100 (Active Treatment) vs Chordate System S200 + CT100 (Placebo Treatment); Test type: Superiority; p = 0.6938, ANCOVA; In the analyses the baseline value was used as a covariate in order to adjust for initial differences at treatment start

2. Secondary Outcome: Change From Baseline in Number of Migraine Days During the 1st, 2nd and 3rd Month and During the Final Four Weeks of the Three Month Post Treatment Investigation Duration
Description: A diary was used where patients added information each day on experienced migraine (yes/no). Baseline was defined as any migraine days from Day -29 until Day -1, i.e. the day before first treatment (Day 1). If the full time period for either baseline or post treatment period was not documented number of migraine days was recalculated with the formula:
  Number of migraine days = (Number of migraine days x 28) / Number of days observed
  If data was missing for any patient for more than 14 days during any period of interest, that patient was excluded from the analysis of that time period.
  The change from baseline in number of migraine days was calculated as follows:
  Change = number of migraine days per four weeks for applicable post treatment period - number of migraine days per four weeks of the baseline period
  As the difference between applicable post treatment period and baseline is presented, negative numbers indicate a post treatment decrease in number of migraine days.
Time Frame: From baseline (28 days pre-treatment) to visit 4 (day 98, ± 7 days)
Population: 44 patients were allocated to active treatment and 43 to placebo. Out of these 40 patients completed the active treatment and 38 patients completed placebo treatment (see participant flow). Only patients who completed treatment were included in analysis. If a patient had missing data for more than 14 days for any of the periods of interest, that period was excluded from the statistical analysis of the applicable endpoint.
Measure: Mean (Standard Deviation); unit: Migraine days/four weeks
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment)
Number analyzed (Participants) | 40 | 38
Migraine days/four weeks
  Month 1 | -1.4 (3.9) | -1.1 (3.9)
  Month 2 | -2.2 (4.0) | -0.8 (3.5)
  Month 3 | -1.4 (4.1) | -2.2 (3.6)
  Final 4 weeks | -1.1 (4.4) | -1.7 (3.3)
Statistical Analysis 1: Comparison: Chordate System S200 + CT100 (Active Treatment) vs Chordate System S200 + CT100 (Placebo Treatment); Null hypothesis: There is no difference between the active treatment and placebo groups in change from baseline in number of migraine days during the 1st month of the three month post treatment investigation duration; Test type: Superiority; p = 0.6557, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Chordate System S200 + CT100 (Active Treatment) vs Chordate System S200 + CT100 (Placebo Treatment); Null hypothesis: There is no difference between the active treatment and placebo groups in change from baseline in number of migraine days during the 2nd month of the three month post treatment investigation duration; Test type: Superiority; p = 0.515, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Chordate System S200 + CT100 (Active Treatment) vs Chordate System S200 + CT100 (Placebo Treatment); Null hypothesis: There is no difference between the active treatment and placebo groups in change from baseline in number of migraine days during the 3rd month of the three month post treatment investigation duration; Test type: Superiority; p = 0.3256, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Chordate System S200 + CT100 (Active Treatment) vs Chordate System S200 + CT100 (Placebo Treatment); Null hypothesis: There is no difference between the active treatment and placebo groups in change from baseline in number of migraine days during the final four weeks of the three month post treatment investigation duration; Test type: Superiority; p = 0.4086, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Responder Rate
Description: "Responder" defined as a patient with 50% or greater decrease in the number of migraine days per four weeks, for the 1st, 2nd and 3rd month post treatment vs baseline
Time Frame: From baseline (28 days pre-treatment) to visit 4 (day 98, ± 7 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment)
Number analyzed (Participants) | 40 | 38
Participants
  Month 1 | 14 | 7
  Month 2 | 15 | 10
  Month 3 | 12 | 15

4. Secondary Outcome: Maximum Migraine Pain Intensity During the 1st, 2nd and 3rd Month, the Final 4 Weeks and the Complete Three Month Post Treatment Investigation Duration
Description: A diary was used where patients added information on the maximum pain intensity on each day according to a 4-point categorical scale (none, mild, medium, severe).
  The maximum documented pain intensity for each patient during each post treatment time period was tabulated for the active treatment and placebo groups.
Time Frame: From baseline (day ≥ - 28 days) to visit 4 (day 98, ± 7 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment)
Number analyzed (Participants) | 39 | 37
Participants
  Month 1: number analyzed (Participants) | 38 | 36
  Month 1: Mild | 6 | 5
  Month 1: Moderate | 13 | 14
  Month 1: Severe | 19 | 17
  Month 2: number analyzed (Participants) | 38 | 36
  Month 2: Mild | 5 | 2
  Month 2: Moderate | 14 | 17
  Month 2: Severe | 19 | 17
  Month 3: number analyzed (Participants) | 36 | 34
  Month 3: Mild | 4 | 8
  Month 3: Moderate | 15 | 14
  Month 3: Severe | 17 | 12
  Final 4 weeks: number analyzed (Participants) | 36 | 34
  Final 4 weeks: Mild | 5 | 5
  Final 4 weeks: Moderate | 18 | 14
  Final 4 weeks: Severe | 13 | 15
  Complete 3 Months: Mild | 1 | 1
  Complete 3 Months: Moderate | 11 | 12
  Complete 3 Months: Severe | 27 | 24

5. Secondary Outcome: Mean Change From Baseline in Median Migraine Duration (Hours/Day) During the 1st, 2nd and 3rd Month, the Final 4 Weeks and the Complete Three Month Post Treatment Investigation Duration
Description: A diary was used where patients added information each day on the number of hours with migraine. The median migraine duration in hours per day was determined for each patient, for each post treatment time period. Baseline for each patient was defined as the median number of migraine hours/day from Day -29 until Day -1, i.e. the day before the first treatment (Day 1).
  The change in median migraine hours/day from baseline, for each defined post treatment time period, was then determined and the mean change is presented.
  As the differences between applicable post treatment period and baseline is presented, negative numbers indicate a post treatment decrease in number of migraine hours/day.
Time Frame: From baseline (28 days pre-treatment) to visit 4 (day 98, ± 7 days)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours / day
Groups:
- Chordate System S200 + CT100 (Active Treatment): Chordate System S200 + CT100 (active treatment): 40 subjects
- Chordate System S200 + CT100 (Placebo Treatment): Chordate System S200 + CT100 (placebo treatment): 38 subjects
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment)
Number analyzed (Participants) | 34 | 32
Hours / day
  Month 1: number analyzed (Participants) | 33 | 30
  Month 1 | -0.7 (3.3) | 0.1 (2.5)
  Month 2: number analyzed (Participants) | 33 | 30
  Month 2 | 0.2 (3.9) | 1.3 (5.0)
  Month 3: number analyzed (Participants) | 31 | 29
  Month 3 | 0.6 (5.1) | -0.4 (4.9)
  Final 4 weeks: number analyzed (Participants) | 31 | 28
  Final 4 weeks | 1.0 (5.7) | 0.0 (4.1)
  Complete 3 Months | -0.6 (3.4) | 0.2 (3.1)

6. Secondary Outcome: Change From Baseline in Drug Consumption for Acute Treatment During the Three Month Post Treatment Investigation Duration
Time Frame: From baseline (28 days pre-treatment) to visit 4 (day 98, ± 7 days)
Population: No statistical analysis was done; only tabular listing. All patients that completed treatment were included.
Measure: Number; unit: Number of medications
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment)
Number analyzed (Participants) | 44 | 43
Number of medications | 157 | 125

7. Secondary Outcome: Patient's Satisfaction as Measured on Clinical Global Impression Scales (CGI)
Description: Patient satisfaction, evaluated by a clinician, was measured using 8-point clinical global impression (CGI) scores on an improvement scale (CGI-I: compared to condition at baseline, how much has changed: 0 = Not assessed, 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse).
Time Frame: At visit 4 day 98, ± 7 days
Population: 44 patients were allocated to active treatment and 43 to placebo. Out of these 40 patients completed the active treatment and 38 patients completed placebo treatment (see participant flow). Only patients who completed treatment were included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment)
Number analyzed (Participants) | 40 | 38
Participants
  Very much improved | 3 | 1
  Much improved | 10 | 5
  Minimally improved | 14 | 12
  No change | 10 | 18
  Minimally worse | 2 | 2
  Much worse | 1 | 0

8. Secondary Outcome: Number of Participants With a Change in Disease-specific Quality of Life From Baseline to End of the Three Month Investigation Duration
Description: Number of Participants with a Change in Disease-specific Quality of Life, as measured by EQ-5D-3L, from Baseline (day 0, visit 2 before first treatment) to End of the Three Month Investigation Duration. EQ-5D-3L uses 5 categorical dimensions - motility, self-care, usual activities, pain/discomfort and anxiety/depression, each classified as improved, no change or worsened.
Time Frame: From baseline (day 0, visit 2) to visit 4 (day 98, ± 7 days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment)
Number analyzed (Participants) | 39 | 38
Participants
  Motility: Improved | 0 | 0
  Motility: No change | 38 | 38
  Motility: Worsened | 1 | 0
  Self-care: Improved | 0 | 0
  Self-care: No change | 39 | 38
  Self-care: Worsened | 0 | 0
  Usual activities: Improved | 0 | 0
  Usual activities: No change | 37 | 37
  Usual activities: Worsened | 2 | 1
  Pain/Discomfort: Improved | 4 | 6
  Pain/Discomfort: No change | 25 | 22
  Pain/Discomfort: Worsened | 10 | 10
  Anxiety/Depression: Improved | 3 | 4
  Anxiety/Depression: No change | 30 | 31
  Anxiety/Depression: Worsened | 6 | 3

9. Secondary Outcome: Disease-specific Quality of Life (VAS Pain Scale) From Baseline to End of the Three Month Study Duration
Description: Disease-specific quality of life, as measured by EQ-VAS, at baseline (day 0, visit 2 before first treatment) and at end of the three month study duration after treatment. The EQ VAS is a standard vertical 20 cm visual analogue scale (similar to a thermometer) for recording an individual's rating for their current health-related quality of life state, with a score from 0-100, where a higher score indicates greater pain intensity.
Time Frame: From baseline (day 0, visit 2) to visit 4 (day 98, ± 7 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment)
Number analyzed (Participants) | 40 | 38
score on a scale
  VAS Pain score at visit 2 | 79.7 (15.0) | 80.6 (15.1)
  VAS pain score at visit 4 | 77.8 (14.5) | 79.8 (15.0)

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected during both the treatment period and the follow-up period until End of Study, an average of 3 months
Arm/Group | Chordate System S200 + CT100 (Active Treatment) | Chordate System S200 + CT100 (Placebo Treatment)
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/43
Other Adverse Events (participants affected / at risk) | 44/44 | 30/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chordate System S200 + CT100 (Active Treatment) (N=44) | Chordate System S200 + CT100 (Placebo Treatment) (N=43)
Laminar hole of the macula (Eye disorders) | 1 (1) | 0 (0) — Pat P7-05 presented with laminar hole of the macula of the right Eye 5 weeks after treatment.The event was assessed as not related to the device and related to the procedure. Conc. diseases were hypertension, dyspepsia and optic neuritis left Eye.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chordate System S200 + CT100 (Active Treatment) (N=44) | Chordate System S200 + CT100 (Placebo Treatment) (N=43)
Increased nasal secretion (Respiratory, thoracic and mediastinal disorders) | 13 | 3
Increased tear secretion (Eye disorders) | 33 | 7
Mild burning sensation (Respiratory, thoracic and mediastinal disorders) | 14 | 3
Paraesthesia of the lip (Respiratory, thoracic and mediastinal disorders) | 14 | 4
Slight discomfort (Respiratory, thoracic and mediastinal disorders) | 23 | 16
Slight pain (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No